CLINICAL TRIAL: NCT04044495
Title: "Sleep, Rhythms and Risk of Alzheimer's Disease: a Daily Life Actigraphic Assessment and MRI Study" "SoRyMA - AMImage3"
Brief Title: Sleep, Rhythms and Risk of Alzheimer's Disease
Acronym: AMImage3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2018/15
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease; Sleep
Keywords: Aging; Sleep/wake Cycle; Hippocampal connectivity; Hippocampal dependant Memory tests; Actigraphy; Functional and structural MRI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample of 100 persons included in AMI / AMImage 2 (Experimental): Sample of 100 persons included in AMI / AMImage 2
  Interventions: Other: Multimodal brain imaging (MRI); Other: Actimetry; Other: Sleep Diary

INTERVENTIONS:
Other: Multimodal brain imaging (MRI) — Multimodal brain imaging (MRI)
Other: Actimetry — 7 days actimetry
Other: Sleep Diary — 7 days Record of sleep and wake cycle

SUMMARY:
Alterations in sleep and the sleep / wake cycle, which are particularly common in Alzheimer's disease patients, could represent an early biomarker for cognitive decline and onset of dementia . Moreover, these disturbances in activity rhythms and sleep patterns represent modifiable factors and therefore potential targets for the prevention of certain neurodegenerative disorders.

The main objective of this study will be to test the hypothesis that elderly people without major cognitive impairment who have circadian rhythm disorders of the sleep / wake cycle have structural and / or functional abnormalities in the central nervous system and more specifically of the hippocampal function which could represent a risk factor for the occurrence of cognitive impairment. Indeed, although many studies in both humans and animals suggest the existence of links between sleep alterations and age-related cognitive impairment, the causality of these observations is still not clear.

This description of the anatomical and functional substratum of sleep / wake cycle alterations occurring in an elderly population will be based on joint analysis of multimodal brain imaging (MRI) and neuropsychology actimetry data. The SoRyMA-AMImage 3 protocol will correspond to the 2nd actimetry measurement point and the 3rd MRI measurement point of a larger population-based cohort AMImage.

This project will collect data from the sleep / wake cycle (actimetry) from a sample of 100 patients included in AMI / AMImage 2 and relate them to brain imaging data (MRI). The main objective of the protocol is the evaluation of the link between changes in sleep and cycle parameters during aging and hippocampal functioning (through fMRI and neuropsychological score of hippocampal dependant tasks). The actimetry variables measured at the two follow-up (4 years apart) will make it possible to measure the degradation of the sleep and cycle parameters (through the reduction of sleep duration, sleep time, increase in sleep fragmentation and decrease in the relative amplitude of the rhythm).

This framework will provide access to a very large amount of data that can be cross-referenced with actimetry data; the longitudinal character of this data collected over a decade will also make it possible to work on the evolution of the actimetry parameters and its relationship with the cognitive and clinical evolution of the subjects. Thus, these data will make it possible to study the prognostic value of the analyzed actimetry parameters in association with very complete clinical and neuropsychological data.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to AMImage 2 cohort and preferentially belonging to subjects included in the first actimetric assessment. AMI subjects have been selected based on Mutualité Sociale Agricole of Gironde (agricultural Health Insurance system database as followed :

  * >65 years old
  * Retired from agriculture
  * Living in Gironde countryside
  * Being affiliated to the French Farmers Health Insurance
* Signed Informed Consent

Exclusion Criteria:

* Left Handed subjects
* Severe dementia (MMSE<13)
* Stroke
* Parkinson's disease
* MRI contraindication
* Health state not allowing displacement to the hospital
* Person under gardianship and not able to give its informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Bold Signal | Day 1
  Bold Signal on Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) Score | Day 1
  seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality
Mannheim Dream questionnaire (MADRE) | Day 1
  MADRE questionnaire evaluates dream recall frequency, emotional aspects of dreams (intensity and tonality), nightmares, lucid dreaming, attitude towards dreams, effects of dreams on waking life and dream literature reading and has been demonstrated to show high retest reliability
Epworth Sleepiness Scale | Day 1
  The test is a list of eight situations in which is rate the tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing
Toronto Alexithymia Scale (TAS-20) | Day 1
  The TAS-20 is a self-report scale that is comprised of 20 items.
  The TAS-20 has 3 subscales:
  * Difficulty Describing Feelings subscale is used to measure difficulty describing emotions. 5 items.
  * Difficulty Identifying Feeling subscale is used to measure difficulty identifying emotions. 7 items.
  * Externally-Oriented Thinking subscale is used to measure the tendency of individuals to focus their attention externally. 8 items.
  Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree.
  The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Positive and Negative Affective Scale (PANAS) | Day 1
  The PANAS Scale or Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire. The test comprises 20 terms, with ten focusing on a positive emotion and the other ten focusing on a negative emotion. The final score of the PANAS Scale / Positive and Negative Affect Schedule (PANAS) test is the sum of the 10 terms on the positive scale and the sum of the 10 terms on the negative scale. The value assigned is positive for answers on the positive scale and negative for answers on the negative scale.
Emotional Regulation Questionnaire (ERQ) | Day 1
  10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores.
Actimetry | Up to 7 days
  Automatically record of waking and sleeping periods on 7 consecutive days
Sleep diary | Up to 7 days
  Series of questions for each 24-hour period with a collection of bedtime, wake-up time, possible night awakenings or even naps

CONTACTS AND LOCATIONS:
Overall Officials: Henri de CLERMONT-GALLERANDE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No